CLINICAL TRIAL: NCT03446976
Title: A Phase 1, Randomized, Open-label, Single-dose, Two-arm, Parallel Group Study to Compare the Pharmacokinetics and Safety of the Pre-filled Syringe and Auto-injector of CT-P13 in Healthy Subjects
Brief Title: CT-P13 (Infliximab) Subcutaneous Administration by Pre-filled Syringe and Auto-injector in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CT-P13 1.9; 135134 (Other: IND)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Health, Subjective

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P13 SC Auto-injector (Experimental): CT-P13 SC Auto-injector
  Interventions: Biological: CT-P13 SC Auto-injector
- CT-P13 SC Pre-filled Syringe (Experimental): CT-P13 SC Pre-filled Syringe
  Interventions: Biological: CT-P13 SC Pre-filled Syringe

INTERVENTIONS:
Biological: CT-P13 SC Auto-injector — Each subject may receive single dose by subcutaneous administration using Auto-Injector
  Arms: CT-P13 SC Auto-injector
Biological: CT-P13 SC Pre-filled Syringe — Each subject may receive single dose by subcutaneous administration using Pre-filled Syringe
  Arms: CT-P13 SC Pre-filled Syringe

SUMMARY:
This study compares two administration methods of CT-P13. Half of participants will receive CT-P13 by pre-filled syringe while the other half will receive CT-P13 by auto-injector.

DETAILED DESCRIPTION:
This is a Phase I Study to Compare Pharmacokinetics and Safety between CT-P13 SC Pre-filled Syringe and CT-P13 SC Auto-injector in Healthy Subjects. A total of 218 healthy subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subject
* Subject voluntarily agrees to participate in this study

Exclusion Criteria:

* Subject with medical history and/or condition
* Female who is pregnant or breastfeeding, or childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
To demonstrate comparable pharmacokinetics (PK) of CT-P13 subcutaneous (SC) administered by auto-injector (AI) versus pre-filled syringe (PFS) in healhty subjects. | over 12 weeks
  Pharmacokinetics will be assessed by AUC

CONTACTS AND LOCATIONS:
Overall Officials: SuEun Song, Study Chair — Celltrion
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No